CLINICAL TRIAL: NCT04146974
Title: Assessing Models of Coordinated Services for Low-Income Children and Their Families
Acronym: AMCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 50685
Record Dates: First submitted 2019-10-14; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Child Development; Family and Household
Keywords: Social services; Coordination; Early childhood education; State and local agencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Assessing Models of Coordinated Services for Low-Income Children and Their Families (AMCS) project is to understand how states and local communities are coordinating services across sectors to most efficiently and effectively serve low-income children and their families. These coordinated services approaches vary along a range of dimensions, including their number and types of partners, funding streams, target populations, goals and objectives, locations, services provided, and monitoring processes. This qualitative study aims to fill gaps in our knowledge by identifying and describing the features of state and local approaches to coordinating early care and education services with family economic security and/or other health and human services.

DETAILED DESCRIPTION:
The purpose of the Assessing Models of Coordinated Services for Low-Income Children and Their Families (AMCS) project is to understand how states and local communities are coordinating services across sectors to most efficiently and effectively serve low-income children and their families. Policymakers and program leaders across the country are experimenting with innovative approaches to combine early care and education, family economic security, and other health and human services (Hulsey et al. 2015; Ross 2018; Sama-Miller and Baumgartner 2017). This qualitative study aims to fill gaps in our knowledge by identifying and describing the features of state and local approaches to coordinating early care and education (ECE) services with family economic security and/or other health and human services.

The AMCS study has six primary research questions:

1. How do state and local coordinated services approaches coordinate partnerships and service application and delivery? What are the experiences of those involved with these coordinated services approaches?
2. How do coordinated services approaches intend to reduce barriers and road blocks for families to access services? Are there federal barriers to implementing such approaches?
3. Are approaches that combine ECE, family economic security, and/or other health and human services able to address other child development factors beyond ECE?
4. What have we learned from efforts to integrate enrollment and eligibility processes for health and human services?
5. Are states and/or localities examining service delivery dynamics across ECE programs to assess availability of care slots and services to meet the needs of eligible families? How are they using data to understand service delivery dynamics?
6. How is public and private ECE funding targeted to meet the needs of at-risk children and families? Are there differences in the families that are able to access services?

The study has three primary ways of collecting information: model profile creation and confirmation for up to 76 coordinated services approaches; telephone interviews with leadership from 20 approaches; and site visits to six coordinated services approaches. Site visits include interviews with staff at the coordinated services approaches and focus groups with parents served by the approach.

The information collected in this study will improve federal, state, and local policymakers', practitioners', and other stakeholders' knowledge and understanding of approaches to coordinating services to support low-income children and their families. Findings will be used to inform the federal government and support their work to set program and evaluation priorities; to inform researchers and others in the field about the state of coordinated services; and finally, to inform practitioners who are currently developing, updating and implementing coordinated services approaches.

ELIGIBILITY:
Inclusion Criteria: Approaches that meet the following criteria are eligible to be included:

* Currently operates in the United States;
* Has a public website or public documents available for review;
* Serves at least some low-income families;
* Directly provides early care and education services for children age 5 and younger;
* Provides family economic security and/or family-focused health and human services in addition to early care and education
* Intentionally coordinates multiple health and human services.

Exclusion Criteria:

* Does not meet in the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Staff and parents from coordinated services approaches serving low-income families and their children.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Features of coordinated services approaches | up to one year
  Study developed template describing components of state and local coordinated services approaches
Qualitative features, service delivery, and perceptions of coordinated services approaches | up to one year
  Telephone interviews (study developed semi-structured telephone interview protocol for state and local coordinated services approaches)
Leader and staff perceptions of coordinated services approaches | up to one year
  Site visits (study developed semi-structured in-person interview protocol with leadership and staff of state and local coordinated services approaches)
Parent/guardian perceptions of coordinated services approaches | up to one year
  Focus groups (study developed semi-structured parent/guardian focus group protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Cavadel, Ph.D., Study Director — Mathematica Policy Research
Locations (1):
- Mathematica, Washington D.C., District of Columbia, United States